CLINICAL TRIAL: NCT04805788
Title: A Phase II Single Arm Trial of Stereotactic Body Proton Radiotherapy (SBPT) for Hepatocellular Carcinoma
Brief Title: Stereotactic Body Proton Radiotherapy for the Treatment of Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200804; NCI-2021-01357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC200804 (Other: Mayo Clinic in Arizona); 20-005638 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-02-24; First posted 2021-03-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Hepatocellular Carcinoma; Stage I Hepatocellular Carcinoma AJCC v8; Stage II Hepatocellular Carcinoma AJCC v8; Stage III Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (SBPT) (Experimental): Patients undergo 1 SBPT fraction over 20-30 minutes per day for a total of 5 fractions.
  Interventions: Radiation: Proton Stereotactic Body Radiation Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Proton Stereotactic Body Radiation Therapy — Undergo SBPT
  Other Names: Proton SBRT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the effect of stereotactic body proton radiotherapy in treating patients with liver cancer. Proton radiotherapy is a type of treatment that uses high-energy beams to treat tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 3-month rate of patients experiencing an increase in Child-Pugh (CP) score by 2 or more points of 5-fraction stereotactic body proton radiotherapy (SBPT) in the treatment of hepatocellular carcinoma (HCC).

SECONDARY OBJECTIVES:

I. To determine the 3-month complication rate as defined by grade 3 or higher acute adverse event.

II. To assess late toxicity with 2 year follow-up. III. To estimate the 6-month local control, liver disease control, progression free survival and overall survival.

IV. To determine objective imaging response rates at 6 months by Modified (m) Response Evaluation Criteria in Solid Tumors (RECIST) and RECIST criteria.

V. To determine the value of volumetric imaging analysis compared to mRECIST and RECIST in the setting of HCC treated with stereotactic body radiotherapy (SBRT).

CORRELATIVE AND EXPLORATORY OBJECTIVES:

I. To evaluate patient-reported outcomes. II. To evaluate clinical features, treatment technique, and dose-volume parameters associated with better local control and fewer adverse events.

III. To determine the value of additional imaging analyses and techniques for assessing tumor response after treatment with SBRT IV. To blood bank patient specimens for future analysis.

OUTLINE:

Patients undergo 1 SBPT fraction over 20-30 minutes per day for a total of 5 fractions.

After completion of study treatment, patients are followed up at 2 weeks, 3 , 6, 12 and 24 months, then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Radiologically presumed or histologically proven, newly diagnosed or recurrent, hepatocellular carcinoma
* Clinical stage T0-T4N0M0 (American Joint Committee on Cancer [AJCC] 8th edition).

  * One to three discrete Liver Reporting and Data System-5 (LIRADS-5) lesions that can be encompassed within a single radiation treatment plan
  * Patients treated with external beam radiation as a bridge to transplant are allowed
  * Minimum single lesion size >= 1 cm, maximum cumulative diameter =< 15 cm
  * Vascular involvement (including portal vein, inferior vena cava [IVC] and/or hepatic vein) is allowed
* Target lesion must be amenable to a SBRT regimen utilizing proton beam therapy (i.e. SBPT)
* Prior local liver treatment including surgery, percutaneous ablation, transarterial bland or chemoembolization (TACE), or Y-90 radioembolization is allowed if completed at least 6 weeks prior to treatment start date
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Life expectance >= 3 months based on medical comorbidities, tumor extent and other clinical factors as determined by treating physician
* Child Pugh score of A or B7
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3 (within 45 days of study entry)
* Platelets (Plt) >= 30,000 cells/mm^3 (the use of transfusion or other intervention to achieve the minimum platelet level is allowed) (within 45 days of study entry)
* Hemoglobin (Hgb) >= 8.0 g/dL (the use of transfusion or other intervention to achieve the minimum hemoglobin level is allowed) (within 45 days of study entry)
* Total bilirubin < 2 mg/dL (within 45 days of study entry)
* Able to and provides Institutional Review Board (IRB) approved study specific written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Enrollment on a second independent protocol is allowed if the second protocol intervention will not significantly affect results of the current protocol as determined by the study investigators

Exclusion Criteria:

* Medical contraindication to receipt of radiotherapy
* Severe active co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or providing informed consent
* Active systemic lupus or scleroderma
* Women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception
* Prior receipt of external beam radiation to the current active disease site or if additional radiotherapy to the current site would be unsafe as determined by the treating radiation oncologist
* More than 3 LIRADS-5 lesions or disease extent such that organ at risk constraints cannot be met
* Tumor extension into common or main branch biliary duct or adjacent organs including stomach, small or large bowel
* Extrahepatic metastases or lymph node involvement
* History of other malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 1 year prior to study entry
* Patient is unable to undergo intravenous contrast enhanced liver imaging (either computed tomography [CT] or magnetic resonance imaging [MRI]) based on clinical imaging protocols established at the treating institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
3-month rate of patients experiencing an increase in Child-Pugh score by 2 or more points of 5-fraction stereotactic body proton radiotherapy in the treatment of hepatocellular carcinoma (HCC) | 3 months
  The rate will be estimated and a 95% exact binomial confidence interval reported, and then tested utilizing a one-sample test for proportions versus the historical control of 15%.

SECONDARY OUTCOMES:
3-month complication rate | 3 months
  Defined by grade 3 or higher acute adverse event. Will be calculated and presented with 95% confidence intervals (CI), while continuous outcomes will be presented with mean, median, 95% CI, and interquartile range (IQR).
Incidence of late toxicity | Up to 2 years
  Defined by grade 3 or higher acute adverse event.
6-month local control | 6 months
  Will be reported via Kaplan-Meier estimates.
Liver disease control | Up to 2 years
  Will be reported via Kaplan-Meier estimates.
Progression free survival | Up to 2 years
  Will be reported via Kaplan-Meier estimates.
Overall survival | Up to 2 years
  Will be reported via Kaplan-Meier estimates.
Imaging response rates | 6 months
  Will be determined by Modified (m) Response Evaluation Criteria in Solid Tumors (RECIST) and RECIST criteria. Will be calculated and presented with 95% CI, while continuous outcomes will be presented with mean, median, 95% CI, and IQR.
Value of volumetric imaging analysis | 6 months
  Will be compared to mRECIST and RECIST in the setting of HCC treated with stereotactic body radiotherapy (SBRT).

OTHER OUTCOMES:
Patient-reported outcomes | Up to 2 years
  Will be evaluated per the validated measure and presented over time with means and 95% CIs.
Clinical features, treatment technique, and dose-volume parameters | Up to 2 years
  Will be associated with better local control and fewer adverse events.
Value of additional imaging analyses and techniques | Up to 2 years
  Will be determined assessing tumor response after treatment with SBRT.
Blood bank patient specimens for future analysis | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B. Ashman, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials